CLINICAL TRIAL: NCT00644709
Title: A Multicenter, Open-Label Extension Study Of High-Risk Hyperlipidemic Patients Treated With An Atorvastatin Starting Dose Adapted To Their Baseline LDL-C Level
Brief Title: A Study Of Atorvastatin For The Treatment Of High Cholesterol In Patients At High Risk Of Coronary Heart Disease (CHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2581112
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin tablets at starting doses of 10, 20, 40, or 80 mg once daily. Three dose adjustments were allowed at baseline, Week 17, and Week 34. Patients who did not meet the LDL-C target at any of these time points had their doses doubled except for those who were on the 80 mg dose. Treatment was given for 52 weeks.

SUMMARY:
A study of the long-term (1 year) effectiveness of atorvastatin to keep patients of high cardiovascular risk at the LDL cholesterol goal of <115 mg/dL

ELIGIBILITY:
Inclusion Criteria:

* Completion of base study
* Dyslipidemia and at high risk of CHD

Exclusion Criteria:

* Impaired liver function
* Gastrointestinal disease that could limit drug absorption

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2003-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Achievement of low-density lipoprotein cholesterol (LDL-C) target of <115 mg/dL | Week 52

SECONDARY OUTCOMES:
Achievement of LDL-C target and total cholesterol target (<190 mg/dL) concomitantly | Week 52
LDL-C, high-density lipoprotein cholesterol (HDL-C), total cholesterol, and triglyceride levels | Baseline and Week 6 for base study; Baseline and Weeks 17, 34, and 52 for extension study
Percent change from baseline of base study in LDL-C, HDL-C, non-HDL-C (triglycerides of >200 mg/dL), total cholesterol, and triglycerides in patients who were statin-naive at baseline of base study | Baseline and Weeks 17, 34, and 52
Achievement of LDL-C target grouped according to whether patients had achieved target at the start of this extension study | Week 52
Adverse events and laboratory test changes | Weeks 17, 34, and 52
Achievement of LDL-C target | Weeks 17 and 34
Achievement of LDL-C target by diabetic patients | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Belgium (15):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brasschaat
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Gilly (charleroi)
  - Pfizer Investigational Site, La Louvière
  - Pfizer Investigational Site, Mechelen
  - Pfizer Investigational Site, Menen
  - Pfizer Investigational Site, Merksem
  - Pfizer Investigational Site, Mortsel
  - Pfizer Investigational Site, Roeselare
  - Pfizer Investigational Site, Seraing
  - Pfizer Investigational Site, Wilrijk
  - Pfizer Investigational Site, Wingene

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581112&StudyName=A%20Study%20Of%20Lipitor%20For%20The%20Treatment%20Of%20High%20Cholesterol%20In%20Patients%20At%20High%20Risk%20Of%20Coronary%20Heart%20Disease%20%28CHD%29